CLINICAL TRIAL: NCT04833608
Title: Using Flexible Carbon Fiber Insoles for 1st Metatarsophalangeal Arthritis Lead to Pain Reduction and High Compliance Rate: A Randomized Controlled Trial
Brief Title: Managing Pain in Patients With MTP Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: VKTRY Gear (Unknown)
Responsible Party: Principal Investigator, Gregory Waryasz, M.D., Orthopaedic Surgeon, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018P002864
Record Dates: First submitted 2021-03-31; First posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-03

CONDITIONS: Hallux Rigidus
Keywords: 1st metatarsophalangeal joint arthritis; 1st MTP arthritis; Hallux Rigidus; foot; Insole; carbon fiber insole; Morton extension insole
MeSH Terms: conditions — Hallux Rigidus

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vktory Carbon fiber insoles (Active Comparator): VKTRY insoles were initially designed to increase ground force leading to a harder push off for faster running or higher jumping. To enable energy return the insole needed to be extremely rigid and therefore consists out of a full length Carbon-Fiber base. Unexpectedly the Carbon fiber base makes this a highly rigid construct which will likely benefit those patients with MTP arthritis as it will take away much movement of the MTP joint, without having an uncomfortable shape, i.e. patients can use this insole in their own shoes, possibly leading to a higher patient compliance and, simultaneously, to better outcome
  Interventions: Device: Vktory insoles
- Morton's extension insoles (Active Comparator): Based on expert opinions, it seems the Morton extensions may alleviate pain but are also poorly tolerated by patients due to its uncomfortable shape, coincidently leading to a low patient compliance rate.
  Interventions: Device: Morton's extension insoles

INTERVENTIONS:
Device: Vktory insoles — Patients were randomized into either the Carbon fiber insole group or Morton's extension group.
  Other Names: Carbon fiber insoles
  Arms: Vktory Carbon fiber insoles
Device: Morton's extension insoles — Patients were randomized into either the Vktory carbon fiber insole group or Morton's extension insole group.
  Arms: Morton's extension insoles

SUMMARY:
Hallux rigidus is a degenerative disease of the first metatarsophalangeal (MTP) joint which affect 2.5% of people over the age of 50. As the arthritis progresses, patients pain levels increase and range of motion decreases. Non-operative management includes the use of NSAIDS, intra-articular injections, shoe modification, activity modifications, and physical therapy. Oral NSAID have been used extensively to reduce swelling and pain but have been found unsatisfactory in providing pain relief. Injections have been shown relieve pain in patients with grade 1 MTP arthritis. Shoe modifications and orthotics can modify the biomechanics of the MTP joint and thereby alleviate pain. Based on expert opinions, it seems the Morton extensions may alleviate pain but are also poorly tolerated by patients due to it's uncomfortable shape, coincidently leading to a low patient compliance rate.

VKTRY insoles were initially designed to increase ground force leading to a harder push off for faster running or higher jumping. To enable energy return the insole needed to be extremely rigid and therefore consists out of a full-length Carbon-Fiber base. Unexpectedly the Carbon fiber base makes this a highly rigid construct which will likely benefit those patients with MTP arthritis as it will take away much movement of the MTP joint, without having an uncomfortable shape, i.e. patients can use this insole in their own shoes, possibly leading to a higher patient compliance and, simultaneously, to better outcome. Even though this insole is being widely used by athletes, no one has explored its role for treating patients with MTP joint arthritis. Therefore, the aim of this study is to compare the VKTRY insole to the current Morton extension insoles in a blinded randomized controlled trial

DETAILED DESCRIPTION:
Subject Enrollment:

Patients were introduced to the study by Foot and Ankle orthopaedic surgeons if they were identified as having hallux rigidis. If the patient agreed, an authorized member of the study staff went through the study in detail and addressed any questions the patients had. If the patient was willing to participate, informed consent was obtained. We emphasized that not participating in the study will not affect their care now or in the future.

Once informed consent was obtained, the patient was randomized into one of two groups.

* Morton Extensions along with current pain management protocol
* VKTRY insoles along with the current pain management protocol

Explanatory variables gathered:

1. Basic patient characteristics
2. Range of motion at 1st MTP joint
3. Hallux Rigidus severity grading

Patients were evaluated at the initial appointment, 2 weeks, 6 weeks, and 12 weeks following their initial appointment. The surveys were given to the patients during each evaluation time point.

Sample Size Calculation:

Based on power analysis to detect a minimal clinically important difference of 10.6 (+/- 4.6 SD) points in the PROMIS pain intensity score between patients using the Vktory carbon fiber insole and patients using Morton's extension insole with an overall two-tailed Type-1 rate of 5%, 80% statistical power and accounting for a 30% lost to follow up, we needed 14 patients in total.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (over 18 years old) with MTP joint arthritis
2. Adults who were competent and able to consent on their behalf
3. Patients who were seen at Massachusetts General Hospital and Newton Wellesley Hospital

Exclusion Criteria:

1. Patients who had history of 1st MTP joint injection
2. Patients that have already used similar orthotics or had prior surgery to the foot
3. Patients who will be treated surgically

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Patient Reported Outcomes Measured Institute System (PROMIS) pain score at 2 weeks, 6 weeks, and 12 weeks | At initial visit, 2 weeks, 6 weeks and 12 weeks
  PROMIS Bank v1.1 pain interference and PROMIS Scale v1.0 pain intensity were completed. Pain Interference instrument measures the self-reported impact of pain on relevant aspects of a person's life and may include the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities. The Pain Intensity instrument is universal rather than disease-specific. The initial items in the Pain Intensity item bank assess pain intensity utilizing a 7-day recall period (items include the phrase "the past 7 days") while the latter item asks patients to rate their pain intensity at the moment.
Change from Baseline Patient Reported Outcomes Measured Institute System (PROMIS) Physical Function at 2 weeks, 6 weeks, and 12 weeks | At initial visit, 2 weeks, 6 weeks and 12 weeks
  PROMIS Bank v2.0 Physical Function was completed. Items included in this reflect mobility, upper limb function (eg, carrying a bag of groceries), and full-body activities (eg, run errands and shop). For the PROMIS measure, the mean T-score in the United States general population is 50 with a SD of 10. Higher scores reflect better physical function.
Change from Baseline Patient Reported Outcomes Measured Institute System (PROMIS) Global Health at 2 weeks, 6 weeks, and 12 weeks | At initial visit, 2 weeks, 6 weeks and 12 weeks
  PROMIS SF v1.1 Global Health was completed. The PROMIS Global health was assessed to understand how patient's symptoms affected physical function, pain, fatigue, emotional distress, social health. The PROMIS global health consists of 10 items with 9 items using five-category response scales, and one item (rating of pain on average) using a response scale of 0-10 that is recoded to five categories.
Change from Baseline Patient Reported Outcomes Measured Institute System (PROMIS) Depression at 2 weeks, 6 weeks, and 12 weeks | At initial visit, 2 weeks, 6 weeks and 12 weeks
  PROMIS Bank v1.0 Depression was completed. The items in the questionnaire focus on the negative moods, emotions, self-image, social cognition and cognitive deficits. A 5-point verbal scale was used to measure patients experience related to their symptoms.
Change from Baseline Compliance and activity Questionnaire at 2 weeks, 6 weeks, and 12 weeks | At initial visit, 2 weeks, 6 weeks and 12 weeks
  Patient compliance was assessed by asking whether the patient used the orthosis - or not. This parameter had two choices that the patient would respond "Yes" or "No" which referred to whether they used the orthosis on the day they completed the questionnaire. Lastly, the comfort rate was measured with a 0-100 Likert scale, where a score of 0 indicated "least comfort" and a score of 100 reflected "best comfort".

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Waryasz, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Newton Wellesley Hospital, Newton, Massachusetts